CLINICAL TRIAL: NCT01976871
Title: A Method to Switch From Oral Dopamine Agonists to Rotigotine in Patients With Restless Legs Syndrome
Brief Title: Switching From Oral Dopamine Agonists to Rotigotine
Acronym: SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: John Winkelman, MD, PhD (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, John Winkelman, MD, PhD, Chief, Sleep Disorders Clinical Research Program, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGH - 2013P000968
Record Dates: First submitted 2013-10-25; First posted 2013-11-06 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Restless Legs Syndrome; Ekbom Syndrome; Willis-Ekbom Disease
Keywords: Restless Legs Syndrome; Ekbom Syndrome; Willis-Ekbom Disease; Rotigotine; Neupro; Dopamine Agonist
MeSH Terms: conditions — Restless Legs Syndrome | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Dopamine Agonist to Rotigotine (Experimental): During the study, we will switch patients who are not satisfied with their current oral dopamine agonist to rotigotine. Cross-titration will allow determination of the lowest effective dose of rotigotine. We will use as initial guidance the equivalence determined from the Parkinson's Disease trials, in which 1 mg rotigotine was shown to be approximately equivalent to 1-1.5 mg ropinirole or 0.25 -0.375 mg pramipexole. Tolerability, adverse events, and RLS symptom control will be evaluated. These data will provide clinicians with practical guidance to optimize RLS treatment while minimizing adverse events.
  Interventions: Drug: Rotigotine

INTERVENTIONS:
Drug: Rotigotine — Rotigotine is FDA approved for the treatment of Restless Legs Syndrome at doses of 1 mg/24h, 2 mg/24h, and 3 mg/24h. The prescribed dose of rotigotine may be achieved using single or multiple patches. Subjects will titrate the dose based on discussions with the investigator.
  Other Names: Neupro

SUMMARY:
The primary objective is to demonstrate safety and tolerability of switching patients with Restless Legs Syndrome (RLS) from an oral dopamine agonist to rotigotine.

As a secondary objective, the investigators will evaluate control of RLS symptoms on rotigotine compared to the prior oral regimen.

DETAILED DESCRIPTION:
The study will consist of 3 in-person visits and 4 scheduled telephone appointments over the course of approximately 6 weeks. The first visit will be the screening visit during which eligibility will be confirmed and informed consent obtained. After the first visit, subjects will continue their current oral dopamine agonist for a one-week baseline period during which they will record RLS symptoms daily.

The second visit will be the baseline visit. The IRLS scale, a commonly used measure of RLS symptoms, will be obtained. An individualized schedule for down-titration of oral dopamine agonist and concomitant up-titration of rotigotine will be provided. After the second visit, subjects will begin this cross-titration. This will entail a pre-determined incremental taper of the oral medication and flexible up-titration of rotigotine according to symptoms. During this time, subjects will keep diaries of RLS symptoms and will speak with the investigator over the phone a total of 3 times (visits 2a-2c) to discuss dosing of rotigotine.

After the titration is complete, subjects will enter the maintenance period, which will last 28 days. There will be another phone contact (2d) one week after the titration is complete to adjust the dose of rotigotine as needed. The subject will then continue the chosen dose for the next 3 weeks of the maintenance period. There will be one final phone contact (2e) 1 week prior to the end of the maintenance period to remind subjects to resume RLS symptom diaries during the final week of the maintenance period.

The third and final visit will take place at the end of the maintenance period. RLS symptoms will be discussed and the IRLS scale, Clinician Global Impression of Change (CGIC), Patient Global Impression of Change (PGIC), and Preference of Medication Scale (POMS) will be administered.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RLS, defined by International Restless Legs Study Group (IRLS) essential criteria:

  1. An urge to move the legs, usually accompanied or caused by uncomfortable and unpleasant sensations in the legs.
  2. The urge to move or unpleasant sensations begin or worsen during periods of rest or inactivity such as lying down or sitting.
  3. The urge to move or unpleasant sensations are partially or totally relieved by movement, such as walking or stretching, at least as long as the activity continues.
  4. The urge to move or unpleasant sensations are worse in the evening or night than during the day or only occur in the evening or night.

(Although some subjects may not meet these criteria on their current oral regimen, these symptoms must have been present prior to treatment.)

* Current treatment with either pramipexole (≤1 mg total daily dose) or ropinirole (≤4 mg total daily dose) with unchanged dose for the past 30 days. Patients also on other RLS medications will be allowed to participate if the dosing has been stable for the past 30 days and the subject agrees to maintain a stable dose for the duration of the trial.
* Inadequate symptom control or patient dissatisfaction with current oral regimen.
* Able to speak and read English.
* Able to provide informed consent.
* Able to learn and demonstrate appropriate patch application.
* Returns appropriately completed RLS symptom log at Visit 2.
* Confirms understanding of cross-titration schedule and is able to restate or summarize these instructions at Visit 2.
* Age ≥18 and ≤75.
* BMI ≥18 and ≤35
* History and/or clinical records document no change in medications active in the central nervous system (antidepressants, analgesics, antipsychotics, antiepileptics, hypnotics, etc.) for at least 30 days prior to visit 1.
* Able to understand study procedures and agrees to remain on stable medications during the period of the study.
* Women of childbearing potential must agree to use a medically accepted method of birth control. Acceptable forms of birth control include:

  1. Condom + spermicide

     * b. Diaphragm + spermicide
     * c. Oral contraceptive pills, hormone implants (like Norplant),or injections (like Depo-Provera)
     * Intrauterine Device

Exclusion Criteria:

* Known secondary cause of RLS, including end-stage renal disease, severe iron deficiency (ferritin <18), pregnancy.
* History of frequent symptomatic orthostatic hypotension.
* Current treatment with a dopamine antagonist medication.
* Another chronic pain syndrome that would, in the opinion of the investigator, interfere with evaluation of RLS symptoms or the response to the study medication.
* Plan to undergo a procedure that may require short or long-term opiates for pain control during the course of the trial.
* Women who are pregnant, lactating, or planning to become pregnant.
* Shift work or other commitments that do not allow for regular sleep at night.
* Known hypersensitivity or intolerance to rotigotine.
* Known allergy to sulfite-containing drugs.
* History of problematic skin hypersensitivity to adhesives.
* Previous or current clinically significant impulse control disorder, as determined by clinical interview.
* Anticipated change in psychiatric or neurologic status likely to require adjustment of CNS-active medications during the study period.
* Unwillingness of subject to remain on stable doses of CNS-active medications.
* Unwillingness of subject to refrain from as-needed use of RLS medications.
* Significant risk for suicide by clinical interview.
* History of severe mental illness or psychosis
* Current unstable medical illness.
* Any medical or psychiatric condition that, in the opinion of the investigator, would interfere with participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Dopamine Agonist to Rotigotine
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oral Dopamine Agonist to Rotigotine
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Completing the Switch and Their Adverse Events
Description: The primary endpoint will be the safety and tolerability of switching from an oral dopamine agonist to rotigotine.
  The CGIC scales were developed to assess treatment outcomes in pharmacological studies. The scales are meant completed by the clinician in person after assessment of the subject. They include 4 global scales describing the severity of illness, change in severity from baseline, therapeutic efficacy, and tolerability of treatment.
  Clinical Global Impression - Improvement scale (CGI-I) rated as: 1, very much improved since the baseline week; 2, much improved; 3, minimally improved; 4, no change from baseline; 5, minimally worse; 6, much worse; or 7, very much worse since the baseline week. The CGI-I was performed at baseline and at Week 5 to see which participants rated as much or very much improved.
  Adverse Events are reported in the Adverse Events module.
Time Frame: Participants will be monitored for the duration of the study, approximately 6-10 weeks depending upon scheduling of visits
Measure: Number; unit: participants
Arm/Group | Oral Dopamine Agonist to Rotigotine
Number analyzed (Participants) | 20
participants
  Oral dopamine agonist to rotigotine switch success | 17
  CGI-I responders (much or very much improved) | 14
  Withdrew due to lack of efficacy | 3

2. Secondary Outcome: International Restless Legs Scale (IRLS)
Description: The IRLS will be used to determine the overall efficacy of RLS symptom control on rotigotine.
  The IRLS is a well-validated instrument for measuring RLS severity during the past week. It includes 10 questions encompassing intensity and frequency of symptoms, associated sleep problems, and the impact of symptoms on the patients' mood and daily functioning. This scale has been shown to have high internal consistency, inter-examiner reliability, test-retest reliability, and convergent validity.
  Minimum score 0, maximum score 40. A decrease in the IRLS score indicates a better outcome.
Time Frame: Study Visit 1 (Day 1) and Study Visit 3 (approximately 35 days after initiating the switch from the oral dopamine agonist to the transdermal rotigotine)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Dopamine Agonist to Rotigotine
Number analyzed (Participants) | 20
units on a scale
  Baseline (Day 1) IRLS score | 19.4 (5.5)
  Week 5 IRLS score | 12.7 (7.7)

3. Secondary Outcome: RLS-6 Scale
Description: The RLS-6 scale will be used to determine the overall efficacy of RLS symptom control on rotigotine, calculated as a mean score for each scale during the final treatment week vs baseline.
  The RLS-6 scale are 11-point (0=not present to 10=very severe) metrics for measuring RLS severity. Four questions delineate a severity profile of RLS during different night and daytime periods: at bedtime, during the night, during the day at rest, during daily activities. The final two questions assess satisfaction with sleep and severity of sleepiness during the day. The RLS-6 scales have been validated on a day-to-day basis, with relatively low placebo effect compared to other RLS rating scales.
  Minimum score 0, maximum score 60. A decrease in the RLS-6 score indicates a better outcome. The RLS-6 scale was completed each day of the study and averaged for the baseline week (approximately days 1-7 of the study) and the final week (approximately days 21-28 of the maintenance period).
Time Frame: Average of Baseline titration week (approximately days 1-7 of the study) vs. Average of Final Treatment week (integrating data from days 28-35 after initiating the switch from the oral dopamine agonist to the transdermal rotigotine)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Dopamine Agonist to Rotigotine
Number analyzed (Participants) | 20
units on a scale
  Baseline RLS symptoms at bedtime | 3.9 (3.2)
  Week 5 RLS symptoms at bedtime | 3.0 (3.1)
  Baseline RLS symptoms during the night | 2.5 (2.3)
  Week 5 RLS symptoms during the night | 2.1 (3.0)
  Baseline RLS symptoms during the day at rest | 2.8 (2.5)
  Week 5 RLS symptoms during the day at rest | 1.4 (2.4)
  Baseline RLS symptoms during daily activities | 1.4 (2.2)
  Week 5 RLS symptoms during daily activities | 0.9 (2.2)

4. Secondary Outcome: Preference of Medication Scale (POM)
Description: The POM will be used to assess patient satisfaction with treatment.
  The POM scale is designed to summarize subjects' preference for the study medication compared to prior therapy. It asks a single question: "How does this current medicine compare to the previous RLS medicine(s) you were taking?" The response set is as follows: (1) Much Better, I prefer this medication (indicating preference for rotigotine); (2) Slightly Better; (3) About the Same; (4) Slightly Worse; (5) Much Worse, I much prefer my previous medication (indicating preference for oral dopamine agonist).
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Oral Dopamine Agonist to Rotigotine
Number analyzed (Participants) | 20
participants
  Much better, I prefer this med | 13
  Slightly better | 2
  About the same | 0
  Slightly worse | 2
  Much worse, I much prefer my previous med | 3

5. Secondary Outcome: The Patient Global Impression of Change Scale
Description: The Patient Global Impression of Change scale (PGIC) will be used to assess patient satisfaction with treatment.
  The PGIC assesses subjective changes in symptoms during clinical trials. This single-item scale asks participants to rate their symptoms as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse." The measure provides a responsive and easily interpretable assessment of participants' evaluations of the importance of their improvement or worsening.
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Oral Dopamine Agonist to Rotigotine
Number analyzed (Participants) | 20
participants
  Very much improved since baseline | 12
  Much improved | 0
  Minimally improved | 3
  No change from baseline | 0
  Minimally worse | 2
  Much worse | 2
  Very much worse since baseline | 1

6. Secondary Outcome: The Clinician Global Impression of Change Scale
Description: The Clinician Global Impression of Change scale (CGIC) will be used to assess patient satisfaction with treatment.
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Oral Dopamine Agonist to Rotigotine
Number analyzed (Participants) | 20
participants
  Very much improved since baseline | 10
  Much improved | 4
  Minimally improved | 1
  No change from baseline | 0
  Minimally worse | 1
  Much worse | 4
  Very much worse since baseline | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Oral Dopamine Agonist to Rotigotine
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 14/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Dopamine Agonist to Rotigotine (N=20)
Somnolence (Nervous system disorders) | 9
Worsening of RLS symptoms during cross-titration (Nervous system disorders) | 6
Skin reaction at patch application site (Skin and subcutaneous tissue disorders) | 5
Insomnia (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 2
Fatigue (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less